CLINICAL TRIAL: NCT01488864
Title: Applied Relaxation for Vasomotor Symptoms in Postmenopausal Women - a Randomized, Controlled Trial
Brief Title: Applied Relaxation for Vasomotor Symptoms
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low drop-out rate and slow recruitment rate
Sponsor: Elizabeth Nedstrand (Other)
Responsible Party: Sponsor-Investigator, Elizabeth Nedstrand, Md, PhD, Ostergotland County Council, Sweden
Organization: Ostergotland County Council, Sweden (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LiÖ/AR-2007
Record Dates: First submitted 2011-12-06; First posted 2011-12-08 (Estimated); Last update posted 2012-05-11 (Estimated); Status verified 2012-05

CONDITIONS: Menopause; Hot Flashes
Keywords: Hot flashes; Vasomotor symptoms; Menopause; Applied Relaxation; Health Related Quality of Life; Salivary cortisol
MeSH Terms: conditions — Hot Flashes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Applied Relaxation (AR) (Experimental)
  Interventions: Behavioral: Applied Relaxation (AR)
- Untreated Control Group (CG) (No Intervention): The women assigned to CG will be told to act as an untreated control group i.e. not to use hormonal treatment, other alternative medication, natural remedies for hot flashes and even not acupuncture, mind-body therapies or intensive physical activity.

INTERVENTIONS:
Behavioral: Applied Relaxation (AR) — AR is a technique influenced on cognitive behavioral therapy using coping mechanism and conditioning. AR focuses on muscle relaxation, where breathing is used for the conditioning of the relaxation. AR implies participation in 10 group sessions during a period of 12 weeks. A therapist will see the women assigned to AR in a group consisted of 6-8 women. The weekly sessions will last for 60 minutes each and are based on a scheme from Öst. The women will be told to practice each component daily.
  During the first session a lecture about menopause and about theories of the mechanisms behind hot flashes will be given.
  The aim of applying AR in view of coping with vasomotor symptoms will be discussed. The group is given a rationale of applying AR as a coping technique for handling sudden unanticipated symptoms by quick calming down, and thus gaining control over the situation.
  Arms: Applied Relaxation (AR)

SUMMARY:
The objectives of this study are to compare frequency and severity of moderate to severe vasomotor symptoms in postmenopausal women treated with applied relaxation (AR) with an untreated control-group (CG) and to investigate if Health Related Quality of Life improve in the AR-group compared to an untreated CG.To study if salivary cortisol excretion would change within the AR treated group compared with the control group.

DETAILED DESCRIPTION:
Approximately 70% of women in Europe and North America experience hot flashes and night sweats during the climacteric period. Many women abstain from hormonal therapy because of side effects or contraindications such as breast cancer or thrombosis.

Different alternative therapies for alleviation of hot flashes are described in the literature. Both pharmacological treatments, different types of natural remedies, acupuncture, life-style changes and mind-body therapies are suggested as promising therapies. Applied relaxation (AR) is a technique influenced on cognitive behavioral therapy (CBT) using coping mechanism and conditioning. Previous study with healthy postmenopausal women showed promising results on hot flash frequency with an average decrease of more than 70 % with persisting effect three months after therapy and also HRQoL significantly increased probably due to better sleep and diminished vasomotor symptoms. But the method must be further investigated before strong evidence-based conclusion can be drawn.

Cortisol is a potent stress hormone regulated by the hypothalamic-pituitary axis. The factors underlying how alternative treatment works and the mechanism underlying improvements in symptoms are not fully understood.

ELIGIBILITY:
Inclusion Criteria:

* postmenopausal women (at least 12 months since last menstrual bleeding occurred or in previously hysterectomised women a serum follicle-stimulating hormone (S-FSH) defined as postmenopausal level according to references at the local laboratory)
* More or equal to 7 moderate to severe hot flashes or more or equal at 50 hot flashes per week according to a two-week screening diary
* ability to understand and speak Swedish
* freely given informed consent

Exclusion Criteria:

* unstable thyroid or other metabolic disease
* treatment with hormone therapy (HT) or other complementary- or alternative treatments treatment for menopausal-related symptoms
* treatment with psychopharmacological drugs and/or sedatives d-un-treated psychiatric disease
* frequently exercising women (≥ 2h high-intensity activities/week)

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2007-03; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Hot flashes average number and severity | Baseline to 12 week after "start of treatment"
  The average number and severity of hot flashes/24 hours in self-registered diaries during the 12th week

SECONDARY OUTCOMES:
Hot flashes | Baseline to 3 months after "end of treatment"
  The average number and severity of hot flashes per 24 hours after 3 months follow-up.
Hot flashes reduction of hot flashes | Baseline to 3 months after "end of treatment"
  The reduction of hot flashes in women defined as responders. Responders are defined as women with ≥50% reduction of hot flashes.
Health Related Quality of Life | Baseline to 3 months "end of treatment"
  The total score in the Women Health Questionnaire measured at 12th week and after 3 months follow-up.
Adverse Events | Baseline to 3 months "end of treatment"
  Adverse events documented by means of using open-ended questions at each contact.
Salivary cortisol | Baseline to 3 months after "end-of-treatment"
  Three samples of salivary cortisol (at awakening, 30 minutes after awakening, and at bedtime)were collected at baseline, after 12 weeks and 3 months after "end-of-treatment"

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Nedstrand, Md, PhD, Principal Investigator — Ostergotland CC, University Hospital Dept. of Obstetrics and Gynecology, 582 85 Linköping, Sweden
Locations (1):
- University Hospital, Dept of Obstetrics and Gynecology, Linköping, Sweden

REFERENCES:
- [Background] Nedstrand E, Wijma K, Lindgren M, Hammar M. The relationship between stress-coping and vasomotor symptoms in postmenopausal women. Maturitas. 1998 Nov 30;31(1):29-34. doi: 10.1016/s0378-5122(98)00058-9. PMID 10091202
- [Background] Nedstrand E, Wijma K, Wyon Y, Hammar M. Applied relaxation and oral estradiol treatment of vasomotor symptoms in postmenopausal women. Maturitas. 2005 Jun 16;51(2):154-62. doi: 10.1016/j.maturitas.2004.05.017. PMID 15917156
- [Background] Nedstrand E, Wijma K, Wyon Y, Hammar M. Vasomotor symptoms decrease in women with breast cancer randomized to treatment with applied relaxation or electro-acupuncture: a preliminary study. Climacteric. 2005 Sep;8(3):243-50. doi: 10.1080/13697130500118050. PMID 16390756
- [Background] Ost LG. Applied relaxation: description of a coping technique and review of controlled studies. Behav Res Ther. 1987;25(5):397-409. doi: 10.1016/0005-7967(87)90017-9. No abstract available. PMID 3318800
- [Background] Hunter MS, Mann E. A cognitive model of menopausal hot flushes and night sweats. J Psychosom Res. 2010 Nov;69(5):491-501. doi: 10.1016/j.jpsychores.2010.04.005. Epub 2010 Jun 1. PMID 20955869
- [Background] Hunter MS, Coventry S, Hamed H, Fentiman I, Grunfeld EA. Evaluation of a group cognitive behavioural intervention for women suffering from menopausal symptoms following breast cancer treatment. Psychooncology. 2009 May;18(5):560-3. doi: 10.1002/pon.1414. PMID 18646246
- [Background] Innes KE, Selfe TK, Vishnu A. Mind-body therapies for menopausal symptoms: a systematic review. Maturitas. 2010 Jun;66(2):135-49. doi: 10.1016/j.maturitas.2010.01.016. Epub 2010 Feb 18. PMID 20167444
- [Background] Vegter S, Kolling P, Toben M, Visser ST, de Jong-van den Berg LT. Replacing hormone therapy--is the decline in prescribing sustained, and are nonhormonal drugs substituted? Menopause. 2009 Mar-Apr;16(2):329-35. doi: 10.1097/gme.0b013e31818c046b. PMID 19188855
- [Background] Hoffmann M, Hammar M, Kjellgren KI, Lindh-Astrand L, Brynhildsen J. Changes in women's attitudes towards and use of hormone therapy after HERS and WHI. Maturitas. 2005 Sep 16;52(1):11-7. doi: 10.1016/j.maturitas.2005.06.003. PMID 16023804
- [Background] Nelson HD, Vesco KK, Haney E, Fu R, Nedrow A, Miller J, Nicolaidis C, Walker M, Humphrey L. Nonhormonal therapies for menopausal hot flashes: systematic review and meta-analysis. JAMA. 2006 May 3;295(17):2057-71. doi: 10.1001/jama.295.17.2057. PMID 16670414
- [Background] Lethaby AE, Brown J, Marjoribanks J, Kronenberg F, Roberts H, Eden J. Phytoestrogens for vasomotor menopausal symptoms. Cochrane Database Syst Rev. 2007 Oct 17;(4):CD001395. doi: 10.1002/14651858.CD001395.pub3. PMID 17943751
- [Background] Wyon Y, Wijma K, Nedstrand E, Hammar M. A comparison of acupuncture and oral estradiol treatment of vasomotor symptoms in postmenopausal women. Climacteric. 2004 Jun;7(2):153-64. doi: 10.1080/13697130410001713814. PMID 15497904
- [Background] Lee MS, Shin BC, Ernst E. Acupuncture for treating menopausal hot flushes: a systematic review. Climacteric. 2009 Feb;12(1):16-25. doi: 10.1080/13697130802566980. PMID 19116803
- [Background] Speroff L, Gass M, Constantine G, Olivier S; Study 315 Investigators. Efficacy and tolerability of desvenlafaxine succinate treatment for menopausal vasomotor symptoms: a randomized controlled trial. Obstet Gynecol. 2008 Jan;111(1):77-87. doi: 10.1097/01.AOG.0000297371.89129.b3. PMID 18165395
- [Background] Wiklund I, Karlberg J, Lindgren R, Sandin K, Mattsson LA. A Swedish version of the Women's Health Questionnaire. A measure of postmenopausal complaints. Acta Obstet Gynecol Scand. 1993 Nov;72(8):648-55. doi: 10.3109/00016349309021159. PMID 8259753
- [Background] Hunter M. The women's health Questionnaire: a meassure of mid-aged women's perceptions on their emotional and physical health. Psycol Health 7: 45-54, 1992
- [Background] Aardal E, Holm AC. Cortisol in saliva--reference ranges and relation to cortisol in serum. Eur J Clin Chem Clin Biochem. 1995 Dec;33(12):927-32. doi: 10.1515/cclm.1995.33.12.927. PMID 8845424
- [Derived] Lindh-Astrand L, Nedstrand E. Effects of applied relaxation on vasomotor symptoms in postmenopausal women: a randomized controlled trial. Menopause. 2013 Apr;20(4):401-8. doi: 10.1097/gme.0b013e318272ce80. PMID 23149867